CLINICAL TRIAL: NCT02850705
Title: The French Cohort and Biobank of Devic's Neuromyelitis Optica and Related Neurological Disorders (NMOSD) (NOMADMUS)
Acronym: NOMADMUS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50742
Record Dates: First submitted 2016-07-22; First posted 2016-08-01 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; Neuromyelitis Optica Spectrum Related Disorders
Keywords: Neuromyelitis Optica; Myelitis; Optic Neuritis; autoantibody; demyelination
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis; Optic Neuritis; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum, CSF, DNA, PBMC
Oversight: Data Monitoring Committee: No

SUMMARY:
Devic's neuromyelitis optica (NMO) is rare. Epidemiological and demographic data are poor, based mainly on monocentric cohorts. Moreover, NMO might be difficult to distinguish from multiple sclerosis and begin with atypical or incomplete clinical presentations. Therefore, NMO is still underdiagnosed. The constitution of a nationwide and prospective cohort, including not only NMO but also clinical syndromes suggestive of a first episode (DNMO-spectrum disorders (SDs)), should allow to gather a critical mass of cases and answer questions that could not have been addressed at the level of a single centre.

Objectives: The main objective is to describe the clinical, radiological and biological features of NMO spectrum disorder (NMO, isolated longitudinally extensive transverse myelitis (LETM), relapsing or not; isolated atypical optic neuritis (ON)) and their evolution. The second aim is to create a biobank dedicated to NMO (serum, whole blood for RNA and DNA extraction, cerebrospinal fluid), to promote translational research in the field. Methods: NOMADMUS is a prospective, multicentre, observational study of patients NMOSD and related disorder in France. Prevalent cases are included retrospectively and then followed prospectively. Incident cases are included from disease onset and followed prospectively. A minimal set of data has been defined and synthesized on specific paper forms derived from the European database for multiple sclerosis (EDMUS) forms. Patients are systematically tested regarding their AQP4-IgG and MOG-IgG status. All the data are centralised in a EDMUS-derived database in Lyon, the EDEN software. All cases are validated and classified by an expert committee.

ELIGIBILITY:
Inclusion Criteria:

Definite Devic's Neuromyelitis Optica NMO according to established criteria (Wingerchuk 1999, Wingerchuk 2006, International panel 2015)

* high risk syndromes for NMOSD, defined as: recurrent or simultaneous optic neuritis, idiopathic single or recurrent longitudinally extensive transverse myelitis (spinal cord lesion seen on MRI >3 vertebral segments)
* patients tested positive for AQP4-IgG autoantibody or MOG-IgG autoantibody
* living in France since 5 years minimum

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Devic's Neuromyelitis Optica NMO
Sampling Method: Non-Probability Sample
Enrollment: 1787 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
number of cases of NMO or NMOSD included in the cohort | At 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon / Hopital Neurologique Pierre Wertheimer, Bron, France

REFERENCES:
- [Derived] Januel E, Brochard V, Le Guennec L, Maillart E, Louapre C, Lubetzki C, Weiss N, Demeret S, Papeix C. Risk factors and prognosis of orotracheal intubation in aquaporin-4-IgG neuromyelitis optica spectrum disorder attacks. Ann Intensive Care. 2024 Jan 8;14(1):4. doi: 10.1186/s13613-023-01213-x. PMID 38185760
- [Derived] Demuth S, Collongues N, Audoin B, Ayrignac X, Bourre B, Ciron J, Cohen M, Deschamps R, Durand-Dubief F, Maillart E, Papeix C, Ruet A, Zephir H, Marignier R, De Seze J; NOMADMUS Study Group. Rituximab De-escalation in Patients With Neuromyelitis Optica Spectrum Disorder. Neurology. 2023 Jul 25;101(4):e438-e450. doi: 10.1212/WNL.0000000000207443. Epub 2023 Jun 8. PMID 37290967